CLINICAL TRIAL: NCT00162461
Title: The Use of Phenytoin Metabolic Ratio as a Putative Marker of CYP2C9 Activity In-vivo
Brief Title: Evaluation of CYP2C9 Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: United States - Israel Binational Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: yc19559-HMO-CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-13 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Phenytoin

ARMS (1):
- Phenytoin (Experimental)
  Interventions: Drug: Phenytoin single dose (300 mg)

INTERVENTIONS:
Drug: Phenytoin single dose (300 mg)

SUMMARY:
The use of phenytoin metabolism to produce S-HPPH accounts for more than 85% of its metabolism. This metabolic pathway is mediated by the activity of CYP2C9.

The purpose of the present study is:

1. To confirm the use of phenytoin metabolic ratio as a marker of CYP2C9 activity
2. To correlate phenytoin metabolic ratio with CYP2C9 genotype
3. To study the frequency distribution of CYP2C9 activity in-vivo

ELIGIBILITY:
Inclusion Criteria:

* Age range of 20-50 years old
* Absence of significant disease states

Exclusion Criteria:

* The presence of significant disease states
* The use of drugs (including birth control pills)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 1998-08; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between phenytoin metabolic ratio and CYP2C9 genotype | 24 hours
Frequency distribution of phenytoin metabolic ratio in the population | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided